CLINICAL TRIAL: NCT04598490
Title: Speed of Premolar Extraction Space Closure: Healed vs Recent Extraction Site- A Prospective Randomized Clinical Trial
Brief Title: Speed of Premolar Extraction Space Closure: Healed vs Recent Extraction Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 53b/2019
Record Dates: First submitted 2020-09-09; First posted 2020-10-22 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Orthodontic Appliance
Keywords: recent; healed; extraction space

STUDY DESIGN:
Intervention Model Description: Space closure into old extraction space
Who Masked: Participant, Outcomes Assessor
Masking Description: After recruiting patients who met the inclusion criteria, the intervention was randomly allocated to either the right or left side using the permuted random block size of 2 with 1:1 allocation ratio. The random sequences for each intervention to either right or left sides was concealed in opaque envelopes and shuffled before the intervention to increase the unpredictability of the random allocation sequence. Each patient was asked to pick a sealed envelope to assign the intervention to either the right or left side. Allocation concealment was aimed to prevent selection bias and to protect the assignment sequence until allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healed extraction site (Experimental): Old Extraction Space
  Interventions: Device: Space closure into old extraction space
- unhealed extraction site (Experimental): Recent Extraction space
  Interventions: Device: Space closure into recent extraction space

INTERVENTIONS:
Device: Space closure into old extraction space — Lower first premolar extraction space was closed using elastic power chain and 0.019X0.025 Stainless steel archwire into healed bony socket
  Arms: Healed extraction site
Device: Space closure into recent extraction space — Lower first premolar extraction space was closed using elastic power chain and 0.019X0.025 Stainless steel archwire into fresh bony socket
  Arms: unhealed extraction site

SUMMARY:
The aim was to compare the rate of teeth movement into fresh and old extraction sites.

DETAILED DESCRIPTION:
Trial design: Randomized controlled clinical trial with a split mouth design. Setting: Jordan University of Science and Technology(JUST) Postgraduate Dental Teaching Clinics and labs.

Participants and interventions: Twenty-eight subjects with bimaxillary proclination requiring extraction of all first premolar teeth participated in this study. In the lower arch, two groups were also identified; group 1 having the first premolar extracted before the commencement of orthodontic treatment and group 2 having the first premolar extracted just before space closure when 0.019 x 0.025 inch SS archwire was reached. Patients were followed-up monthly for three months. At every follow-up visit lower alginate impressions were taken. Extraction spaces in the lower arch follow-up models were measured using digital caliper.

The rate of extraction space closure in the lower arch was assessed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Proclined upper and lower incisors (Ui/max >115 o, Li/mand >99o)
* Mild upper and lower arch crowding (<4mm) or no crowding
* Need for upper and lower first premolars extraction
* Skeletal I malocclusion (1<ANB <5)
* Average lower facial height and maxillomandibular plane angle (22 o <MM<32 o)
* Class I canine relationship
* Good oral hygiene and healthy periodontium

Exclusion Criteria:

* Poor oral hygiene
* Diseases and medications that were likely to affect bone biology
* Previous orthodontic treatment
* Evidence of bone loss
* Active periodontal disease
* Smoking

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Amount of space closure | 3 months
  Width of extraction space will be measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Elham S A Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Faculty of Dentistry/Jordan University of Science and Technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No